CLINICAL TRIAL: NCT00755651
Title: Studies on the H Pipelle, a New Device for Endometrial Sampling at Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Free Hampstead NHS Trust (Other)
Responsible Party: Adam Magos BSc MB BS MD FRCOG, Consultant Gynaecologist, Royal Free Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: REC 6056
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Abnormal Uterine Bleeding
Keywords: Menorrhagia; Uterine fibroids; Endometrial polyps; Endometrial cancer
MeSH Terms: conditions — Metrorrhagia; Menorrhagia; Leiomyoma; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- H Pipelle (Experimental): Endometrial sample obtained using the H Pipelle
  Interventions: Procedure: Endometrial biopsy
- Pipelle (Active Comparator): Endometrial sample obtained with standard Pipelle
  Interventions: Procedure: Endometrial biopsy

INTERVENTIONS:
Procedure: Endometrial biopsy — Endometrial biopsy taken on completion of office/outpatient diagnostic hysteroscopy
  Other Names: Pipelle; H Pipelle

SUMMARY:
The investigators have developed a novel instrument for taking endometrial biopsies at no touch (vaginoscopic) hysterectomy which avoids the need to instrument the vagina with speculums and tenaculums, and also avoids the possible need for cervical dilatation. The investigators wish to study the ease of use and efficacy of the new device compared with traditional techniques of endometrial sampling at hysteroscopy.

DETAILED DESCRIPTION:
We have developed a novel instrument for taking endometrial biopsies at no touch (vaginoscopic) hysterectomy which avoids the need to instrument the vagina with speculums and tenaculums, and also avoids the possible need for cervical dilatation. We wish to study the ease of use and efficacy of the new device compared with traditional techniques of endometrial sampling at hysteroscopy in terms of biopsy adequacy, the time taken to obtain a biopsy and patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Indication to carry out diagnostic hysteroscopy
* Agrees and is suitable for outpatient/office hysteroscopy

Exclusion Criteria:

* Failed outpatient/office hysteroscopy

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2003-01; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Discomfort | End of procedure

SECONDARY OUTCOMES:
Procedure time, biopsy adequacy | End of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Adam Magos, BSc MD FRCOG, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (1):
- Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Result] Sharma M, Taylor A, di Spiezio Sardo A, Buck L, Mastrogamvrakis G, Kosmas I, Tsirkas P, Magos A. Outpatient hysteroscopy: traditional versus the 'no-touch' technique. BJOG. 2005 Jul;112(7):963-7. doi: 10.1111/j.1471-0528.2005.00425.x. PMID 15958000